CLINICAL TRIAL: NCT06416891
Title: Effect of Adding Dexamethasone to Bupivacaine 0.25% in Superficial Cervical Plexus Block on Surgical Field Visibility During Tympanomastoid Surgery in Adults, A Randomized Controlled Study
Brief Title: Effect of Adding Dexamethasone to Bupivacaine 0.25% in SCPB on Surgical Field Visibility During Tympanomastoid Surgery
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Kareem Mohammed Assem Nawwar, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MS-426-2023
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Surgical Field; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bupivacaine (Active Comparator): SCPB will be administered using 10 ml of bupivacaine 0.25% (5 ml of bupivacaine 0.5% + 5 ml of normal saline).
  Interventions: Drug: bupivacaine 0.25%
- Bupivacaine plus dexamethasone (Active Comparator): SCPB will be administered using dexamethasone 2 mg in 10 ml of bupivacaine 0.25% (5 ml of bupivacaine 0.5% + dexamethasone 0.5 ml + 4.5 ml of normal saline).
  Interventions: Drug: dexamethasone 2 mg in bupivacaine 0.25%

INTERVENTIONS:
Drug: bupivacaine 0.25% — SCPB using 10 ml of bupivacaine 0.25%
  Arms: Bupivacaine
Drug: dexamethasone 2 mg in bupivacaine 0.25% — SCPB using dexamethasone 2 mg in 10 ml of bupivacaine 0.25%
  Arms: Bupivacaine plus dexamethasone

SUMMARY:
The aim of this study is to evaluate the efficacy of adding dexamethasone to bupivacaine 0.25% in ultrasound-guided SCPB on surgical field visibility during tympanomastoid surgery.

DETAILED DESCRIPTION:
Tympanomastoid surgery is a commonly performed otological procedure performed to treat various middle ear pathologies, including chronic otitis media, cholesteatoma, and mastoiditis (1). One of the most significant complications associated with tympanomastoid surgery is bleeding, which can result in surgical difficulties, prolonged operative time, and increased morbidity (2).

Pain is also a major concern post-surgery and can lead to patient discomfort and dissatisfaction (3). Achieving optimal surgical field visibility is of paramount importance to ensure precise and safe surgical interventions. However, the presence of intraoperative bleeding and inadequate visualization can significantly impede the surgeon's ability to perform the procedure effectively, leading to potential complications and suboptimal outcomes (4).

Conventional methods for pain management during tympanomastoid surgery often involve general anesthesia or local infiltration of anesthetic agents around the surgical site. However, these techniques may not adequately address pain control and can be associated with unwanted systemic side effects (5).

To minimize bleeding and pain and improve surgical field visualization, anesthetic techniques such as induced hypotension have been used to achieve adequate homeostasis and surgical field visualization during surgery (4).

Induced hypotension involves reducing systemic blood pressure, thereby decreasing blood flow to the surgical site, minimizing the risk of bleeding, and improving the surgical field's visualization, leading to better surgical outcomes (5). However, induced hypotension can lead to cerebral hypoperfusion, organ damage, and other serious complications (6).

The use of regional anesthesia techniques, such as ultrasound-guided superficial cervical plexus block (SCPB), has gained considerable attention as a potential adjunct to general anesthesia (7). SCPB block involves the deposition of local anesthetic agents around the superficial cervical plexus, which provides sensory innervation to the ear, mastoid, and surrounding structures (8).

The SCPB provides effective analgesia and reduces sympathetic activity, resulting in reduced bleeding and improved surgical conditions (9). Also, the superficial cervical plexus provides sensory innervation to the ear and surrounding structures, reducing pain perception during and after surgery (10).

Modern medicine focuses on enhancing patient outcomes and reducing surgical complications through improved surgical field visualization. Advanced imaging technologies like intraoperative MRI or CT scanners offer real-time, high-resolution images, aiding accurate tumor localization (11). Fluorescence-guided agents like indocyanine green enhance visualization of blood vessels, lymph nodes, and tumors during surgery. Augmented reality (AR) and virtual reality (VR) systems provide valuable guidance, allowing surgeons to identify critical structures, plan optimal incisions, and simulate complex procedures pre-surgery. Robot-assisted surgery offers enhanced precision and 3D visualization through high-definition cameras. These combined methods lead to safer and more effective surgical interventions (12).

Recent studies have suggested that combining bupivacaine, a long-acting local anesthetic, with dexamethasone, a potent anti-inflammatory agent, may offer several advantages (13). Bupivacaine provides prolonged pain relief, while dexamethasone reduces local inflammation and edema, potentially improving surgical field visibility (14).

To our knowledge, this is the first randomized clinical trial investigating the effect of adding dexamethasone to bupivacaine 0.25% in ultrasound-guided SCPB on surgical field visibility during tympanomastoid surgery in adults.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I & ASA II patients
2. Patients undergoing tympanomastoid surgery.
3. Age group: from 21 to 70 years old.
4. Duration of surgery less than 5 hours.

Exclusion Criteria:

* Patient refusal.
* Uncooperative patients.
* Allergy to local anesthetics or dexamethasone.
* Anatomical abnormalities include malformations, deformities, growths, or structural irregularities.
* Infection at injection site.
* Coagulopathy: PTT > 40 seconds, INR > 1.4, platelet count < 100x10⁹. or drug induced bleeding disorders

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Modena bleeding score | up to 5 hours
  Grading of surgical field visualization

SECONDARY OUTCOMES:
Surgeon satisfaction | 1 hour postoperatively
  Scoring surgeon satisfaction with the 3-point scale (1: good, 2: sufficient, 3: unfavorable)
Analgesia duration | 24 hours
  Time to first call for a rescue analgesic
Postoperative pain | 24 hours postoperatively
  Postoperative pain is measured by Visual Analog Scale (0 = no pain, 10 = worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Sahar MM El-Shall, M.D., Study Chair — Professor of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Mohsen M Waheb, M.D., Study Director — Lecturer of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Kareem MA Nawwar, M.D., Study Director — Lecturer of Anesthesiology, Surgical ICU & Pain Management, Cairo University; Aboumazen A Abouhashem, M.B.B.Ch., Principal Investigator — Resident of Anesthesia, Surgical ICU & Pain Management
Locations (1):
- Faculty of Medicine, Cairo University, Cairo, Egypt